CLINICAL TRIAL: NCT03108898
Title: Progenitor Cells in Human Esophagus
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dennis Wigle, MD, PhD, Mayo Clinic
Other Study IDs: 17-000700
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Progenitor Cells; Aging, Cells; Esophagus Disorder
MeSH Terms: conditions — Esophageal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Esophageal tissue will be collected at the time of the patient's surgery in excess of clinical diagnosis (i.e. tissue that would otherwise be discarded). The researchers will analyze sections of adult esophagus tissue for the presence of CD34+ sox2+ progenitor cells to determine the number of progenitors present at a particular age of patient. The researchers will also examine sections of different portions of the esophagus, to determine whether certain sections contain more progenitors, and thus perhaps a greater ability to regenerate, than others.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to better understand how esophageal cells change with age.

DETAILED DESCRIPTION:
The researchers will collect information from the patient's medical record and collect esophageal tissue at the time of the patient's surgery in excess of clinical diagnosis (i.e. tissue that would otherwise be discarded). There will be no patient contact after the patient's surgery. The researchers will analyze sections of adult esophagus tissue for the presence of CD34+ sox2+ progenitor cells to determine the number of progenitors present at a particular age. The researchers will also examine sections of different portions of the esophagus, to determine whether certain sections contain more progenitors, and thus perhaps a greater ability to regenerate, than others.

This study involves testing DNA and patients will not be notified of the genetic test results and the results will not be put into their medical record. Patients will be asked to give consent to have any remaining esophageal tissue used for future studies of esophageal disease at Mayo Clinic, learn about, prevent, or treat any other health problems and give their sample and related information to researchers at other institutions.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Esophagus surgery at Mayo Clinic

Exclusion Criteria:

* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing esophageal surgery at Mayo Clinic Rochester
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Amount of Progenitor Cells | 1 year
  We will examine sections of different portions of the esophagus, to determine whether certain sections contain more progenitors, and thus perhaps a greater ability to regenerate, than others.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials